CLINICAL TRIAL: NCT00176891
Title: Phase II Study of Combined Laronidase (AldurazymeTM) Enzyme Replacement Therapy (ERT) With Hematopoietic Stem Cell Transplantation (HSCT) for Hurler Syndrome (MPS IH)
Brief Title: Stem Cell Transplant w/Laronidase for Hurler
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Masonic Cancer Center, University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MT2004-09; 0403M57728 (Other: IRB, University of Minnesota)
Record Dates: First submitted 2005-09-12; First posted 2005-09-15 (Estimated); Results first posted 2019-07-11 (Actual); Last update posted 2019-07-11 (Actual); Status verified 2019-07

CONDITIONS: Mucopolysaccharidosis I; Hurler Syndrome
Keywords: Laronidase ERT; Stem cell transplant; storage disease; inborn errors of metabolism; hurler syndrome; glycosaminoglycans; enzyme replacement
MeSH Terms: conditions — Mucopolysaccharidosis I; Metabolism, Inborn Errors | interventions — Stem Cell Transplantation; Iduronidase

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Laronidase ERT Treatment (Experimental): Weekly infusion of laronidase enzyme replacement therapy followed by hematopoietic stem cell transplant.
  Interventions: Procedure: Stem Cell Transplant; Drug: Laronidase ERT

INTERVENTIONS:
Procedure: Stem Cell Transplant — enzyme replacement 10-12 weeks prior to hematopoietic stem cell transplant (HSCT), and 8 weeks following
  Other Names: ERT
Drug: Laronidase ERT — Laronidase ERT will be administered 10-12 weeks prior to HSCT, and 8 weeks following.
  Other Names: Aldurazyme®

SUMMARY:
The investigators hypothesize that weekly infusions of Laronidase ERT for 10-12 weeks prior to transplant and 8 weeks following transplant will result in a reduction of glycosaminoglycans (GAG) burden that is associated with decreased complications following transplant.

DETAILED DESCRIPTION:
Subjects will receive laronidase once a week intravenously for 10-12 weeks prior to transplant and for approximately 8 weeks after transplant. Laronidase will be given by intravenous infusion (IV) through a catheter and from there to your child's body's cells and organs to break down the glycosaminoglycans (GAG) buildup.

Prior to starting ERT, subjects will have a complete physical examination, which includes a complete assessment of your child's airway and lungs. In addition to standard treatment evaluations and tests, which are done prior to hematopoietic stem cell transplant (HSCT), subjects will have the following tests: an additional teaspoon of blood for a baseline test for serum antibodies against laronidase, before and after the fourth dose of laronidase, the investigators will collect 2 teaspoons of blood for an alpha-L-iduronidase enzyme level; to watch for side effects to laronidase and the development of antibodies to laronidase, approximately 2 teaspoons of blood will be collected every 3 weeks while the subject is receiving laronidase ERT.

ELIGIBILITY:
Inclusion Criteria:

* Patients with the diagnosis of mucopolysaccharidosis type IH (MPS I, Hurler syndrome) who are candidates for first hematopoietic stem cell transplant (HSCT) according to a University of Minnesota myeloablative HSCT protocol.

Exclusion Criteria:

* Not being considered for University of Minnesota myeloablative HSCT protocol.
* Previous administration of laronidase enzyme
* Second or subsequent HSCT.

Max Age: 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 25 (Actual)
Dates: Start 2004-03; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paul Orchard, MD, Principal Investigator — Masonic Cancer Center, University of Minnesota
Locations (1):
- Masonic Cancer Center, University of Minnesota, Minneapolis, Minnesota, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Laronidase ERT Treatment
Started | 25
Completed | 22
Not Completed | 3

BASELINE CHARACTERISTICS:
Arm/Group | Laronidase ERT Treatment
Number analyzed (Participants) | 22
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 22
  Between 18 and 65 years | 0
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 11
Region of Enrollment [Number; unit: participants]
  United States | 22

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients Alive at One Year Post Transplant
Time Frame: one year
Measure: Count of Participants; unit: Participants
Arm/Group | Laronidase ERT Treatment
Number analyzed (Participants) | 22
Participants | 18

2. Primary Outcome: Number of Patients Requiring Ventilator Support at One Year Post Transplant
Time Frame: one year
Measure: Count of Participants; unit: Participants
Arm/Group | Laronidase ERT Treatment
Number analyzed (Participants) | 22
Participants | 6

3. Secondary Outcome: Donor Engraftment
Time Frame: Day 100 post transplant
Measure: Count of Participants; unit: Participants
Arm/Group | Laronidase ERT Treatment
Number analyzed (Participants) | 22
Participants | 21

4. Secondary Outcome: Patients With Grade III-IV Acute GVHD
Time Frame: Day 100 post transplant
Measure: Count of Participants; unit: Participants
Arm/Group | Laronidase ERT Treatment
Number analyzed (Participants) | 22
Participants | 1

5. Secondary Outcome: Reduction in Glycosaminoglycans (GAG)
Description: Data was not collected on this outcome measure and is not available for reporting.
Time Frame: Prior to, During and After ERT
Population: Data was not collected on this outcome measure and is not available for reporting.
Arm/Group | Laronidase ERT Treatment
Number analyzed (Participants) | 0

6. Secondary Outcome: Toxicity (Adverse Events) Associated With Infusions of Laronidase
Description: Data was not collected on this outcome measure and is not available for reporting.
Time Frame: 1 year post transplant
Population: Data was not collected on this outcome measure and is not available for reporting.
Arm/Group | Laronidase ERT Treatment
Number analyzed (Participants) | 0

7. Secondary Outcome: Development of Anti-iduronidase Antibodies in Serum
Time Frame: 1 Year
Population: Data was not collected on this outcome measure and is not available for reporting.
Arm/Group | Laronidase ERT Treatment
Number analyzed (Participants) | 0

8. Secondary Outcome: Patients With Improvement in Obstructive Apnea (Breathing) by Polysomnography
Time Frame: Baseline, 12 weeks after laronidase, after transplant
Population: Data was not collected on this outcome measure and is not available for reporting.
Arm/Group | Laronidase ERT Treatment
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Description: An SAE as defined by the protocol includes unexpected: 1) laronidase related toxicity which is life threatening, requires hospitalization, causes persistent or significant disability/incapacity, causes congenital anomaly, is a medical event that may jeopardize the patent and require medical/surgical intervention to prevent one of the other outcomes, or causes death; 2) graft failure; 3) severe acute GVHD; and 4) severe regimen related toxicity grade III-IV, which includes mortality.
Arm/Group | Laronidase ERT Treatment
Serious Adverse Events (participants affected / at risk) | 6/22
Other Adverse Events (participants affected / at risk) | 21/22
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Laronidase ERT Treatment (N=22)
Heart failure (Cardiac disorders) | 1
Pericardial effusion (Cardiac disorders) | 1
Multiple system organ failure (General disorders) | 1
Other, Infection NOS (Infections and infestations) | 2
Catheter-related infection (Infections and infestations) | 1
Other, Upper respiratory Tract infection (Infections and infestations) | 1
Multifocal cerebral infarct (Nervous system disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Laronidase ERT Treatment (N=22)
Increased Liver Function Test (Hepatobiliary disorders) | 1
Acute Respiratory Distress (Respiratory, thoracic and mediastinal disorders) | 1
Hyperbilirubinemia (Hepatobiliary disorders) | 1
Blood/Bone Marrow, NOS (Blood and lymphatic system disorders) | 2
Cerebrovascular Ischemia (Nervous system disorders) | 1
Cardiac, NOS (Cardiac disorders) | 1
Cholecystitis (Hepatobiliary disorders) | 1
Dehydration (Gastrointestinal disorders) | 1
Diarrhea (Gastrointestinal disorders) | 4
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1
Fatigue (General disorders) | 1
Fracture, NOS (Musculoskeletal and connective tissue disorders) | 1
Hypoglycemia (Metabolism and nutrition disorders) | 1
Hemoglobin, NOS (Blood and lymphatic system disorders) | 1
Hemolysis (Blood and lymphatic system disorders) | 1
Hemorrhage, Pulmonary (Respiratory, thoracic and mediastinal disorders) | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2
Infection with Grade 3 or 4 Neutrophils (Infections and infestations) | 1
Infection, NOS (Infections and infestations) | 3
Infection with Normal Neutrophils (Infections and infestations) | 1
Infection with Unknown Neutrophils (Infections and infestations) | 13
Mucositis, Pharynx (Respiratory, thoracic and mediastinal disorders) | 1
Necrosis, GI (Gastrointestinal disorders) | 1
Neurology, NOS (Nervous system disorders) | 1
Obstruction, Ureter (Renal and urinary disorders) | 1
Pain, Abdomen (Gastrointestinal disorders) | 2
Pain, Cardiac (Cardiac disorders) | 1
Pulmonary, NOS (Respiratory, thoracic and mediastinal disorders) | 2
Rash/Desquamation (Skin and subcutaneous tissue disorders) | 1
Renal, NOS (Renal and urinary disorders) | 1
Supraventricular and Nodal Arrythmia (Cardiac disorders) | 1
Syncope (Nervous system disorders) | 1
Thrombosis (Vascular disorders) | 2
Vascular, NOS (Vascular disorders) | 1

LIMITATIONS AND CAVEATS:
All of the patients on this trial also underwent allogeneic blood/marrow transplantation. All the serious and non-serious adverse events listed were related to the process of transplantation and not to the study medication, Laronidase.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No